CLINICAL TRIAL: NCT02407340
Title: Laboratory Studies on Oxytocin for Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00033324
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Alcoholism; Alcohol Related Disorders
Keywords: Alcohol Withdrawal Delirium
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Alcohol Withdrawal Delirium | interventions — Oxytocin; Benzyl Alcohols

STUDY DESIGN:
Intervention Model Description: Oxytocin vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): intranasal oxytocin - 40 International Units (IU) dose administered 3 times daily for 1 week
  Interventions: Drug: oxytocin
- Placebo (Placebo Comparator): Intranasal placebo administered 3 times daily for 1 week
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxytocin — 40 international Units (IU) 3xday delivered as 5 sprays (0.1 mL) per nostril
  Other Names: syntocinon
  Arms: Oxytocin
Drug: placebo — 5 sprays (0.1 mL) per nostril 3xday; bottles are identical to those of active drug
  Other Names: (Na Cl 0.65%, Phenylcarbinol, Benzalkonium Cl)
  Arms: Placebo

SUMMARY:
This study will examine the utility of the neuropeptide oxytocin (OT) as a potential new medication for the treatment of Alcohol use disorder (AUD). Non-treatment seeking men and women with AUD will be enrolled in a double blind placebo controlled phase I clinical trial. Participants will complete an 7-day inpatient protocol. During the first 3 days of the inpatient protocol, participants will complete alcohol abstinence in which withdrawal symptoms are measured,and urine will be collected to determine withdrawal symptom severity and urine levels of the stress hormone cortisol. Participants will then complete 3 laboratory procedures which measure 1) stress response, 2) motivation to drink alcohol and 3) subjective and physiological effects of alcohol. Finally, because participants are individuals with AUD, investigators will administer a brief intervention to address their risky alcohol drinking and problems before discharge.

DETAILED DESCRIPTION:
This study will lay the necessary groundwork for future comprehensive research to examine the utility of the neuropeptide oxytocin (OT) as a potential new medication for the treatment of Alcohol use disorder (AUD). OT modulates a number of key systems involved in addiction processes, including dopamine (DA) mesolimbic reward circuitry, and hypothalamic-pituitary-adrenal (HPA) axis and corticotrophin-releasing factor (CRF) stress systems, and has low abuse liability. Our overarching hypothesis is that OT will attenuate several measures thought to drive compulsive alcohol drinking and relapse. Specifically, investigators will examine whether OT decreases acute stress responses, alleviates alcohol withdrawal symptoms, reduces craving and motivation to drink, and decreases alcohol self-administration. Since interactions with alcohol are an important focus of our study, investigators will enroll non-treatment seeking heavy drinkers with AUD in a double blind, placebo controlled inpatient protocol. Subjects will be randomized to receive intranasal OT (40 IU/dose) or placebo 3 times daily. Participants will complete alcohol detoxification; investigators will measure alcohol withdrawal symptoms, craving, and 24-hr urinary free CORT. Participants will then complete 3 laboratory procedures in fixed order. The Trier Social Stress Test (TSST) which includes public speaking and performance of mental arithmetic will be used to examine subjective and physiological stress responses. An alcohol motivated responding (AMR) procedure will be used to examine subjects' responding to earn either drinks or money. A cumulative alcohol-dosing (CAD) procedure will be used to examine physiological and subjective responses across several blood alcohol levels. cortisol (CORT) levels will also be assessed. This study will provide new information on OT efficacy across a range of different measures predictive of alcohol use and misuse, and, if OT shows efficacy, help clarify the mechanism of OT action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 21-50 years old male and female subjects
* Must meet Diagnostic and Statistical Manual (DSM) -V criteria for AUD and not be seeking treatment
* Actively drinking
* Positive blood phosphatidylethanol (PEth) blood test

Exclusion Criteria:

* Current DSM-V major current mood or anxiety disorder or drug use disorder (excluding alcohol and nicotine use disorders, and moderate-severe cannabis use disorder); in or in need of treatment
* Drug use in last 30 days and/or positive urine toxicology screens (excluding marijuana)
* History of seizure disorder or closed head trauma
* History of withdrawal-related seizures or serious alcohol withdrawal symptoms
* HIV positive
* Neuroendocrine disorder
* Any serious medical condition that would place subject at risk or interfere with study participation
* Liver function tests more than 3 times normal at screening
* Prescription medications in last 3 months that could affect central nervous system or HPA axis function
* Women who are pregnant, nursing or planning pregnancy cannot participate

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Alcohol drinking | 1 day
  Group mean number of Standard Drink Units earned and self-administered in the laboratory session

SECONDARY OUTCOMES:
alcohol effects | 1 day
  Group mean stimulation and sedation subscale scores on the biphasic alcohol effects scale (BAES), a 14-item scale consisting of adjectives that describe the stimulant- and sedative-like effects of alcohol. The items are presented in alphabetical order, and are rated on an 11-point rating scale from 0=Not at All to 10=Extremely after controlled alcohol administration.
side effects | 1 week
  side effects reported on the Systematic Assessment for Treatment Emergent Events (SAFTEE)
Salivary cortisol | 1 day
  Peak and Area under the curve salivary cortisol levels after trier social stress test

CONTACTS AND LOCATIONS:
Overall Officials: Elise Weerts, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

DOCUMENTS (1):
  • Study Protocol (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT02407340/Prot_000.pdf